CLINICAL TRIAL: NCT07238439
Title: Scenario-Driven Virtual Reality Game for Dementia Education Among Healthcare Students: Protocol for a Four-Arm Study
Brief Title: Scenario-Driven Virtual Reality Game for Dementia Education Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Chiba University (Other); Tokyo University (Other)
Responsible Party: Principal Investigator, Dianis Wulan Sari, Principal Investigator, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3759-KEPK
Record Dates: First submitted 2025-09-20; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Dementia
Keywords: Aged; Dementia; Education program; Healthcare student; Long-term care; Virtual reality
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Participants in this study were drawn from a previous study (NCT06629844), which employed a quasi-experimental, two-arm design. In the current study, each of the two groups from the previous study (intervention and control) was further divided into two subgroups, resulting in a total of four groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR-Experienced + ASA VR Group (Experimental): This arm includes participants who have previously engaged with a VR-based dementia education program. For this study, they will receive the full intervention, which combines the ASA VR content.
  Purpose: This group helps assess the incremental benefit of the ASA content when integrated with prior VR exposure, evaluating how additional structured content enhances existing VR learning.
  Interventions: Other: VR-Experienced + ASA VR Group
- VR-Experienced + Standard Control Group (Active Comparator): This arm consists of participants who have also previously engaged with a VR-based dementia education program. However, for this study, they will only receive the standard course material on dementia through the university's e-learning platform. They will not receive any ASA VR exposure.
  Purpose: This group serves as a comparison to Arm 1, helping to isolate the specific impact of the ASA VR intervention for those with prior VR experience, by observing outcomes when no further structured intervention is provided beyond the regular curriculum.
  Interventions: Other: VR-Experienced + Standard Control Group
- VR-Unexposed + ASA VR Group (Experimental): This arm comprises participants who have no prior exposure to a VR-based dementia education program. For this study, they will receive the full intervention, combining the immersive ASA VR content.
  Purpose: This group allows for a direct assessment of the overall effectiveness of the complete ASA VR program for students new to this type of intervention, comparing it against conventional learning for a previously unexposed group.
  Interventions: Other: VR-Unexposed + ASA VR Group
- VR-Unexposed + Standard Control Group (Active Comparator): This arm includes participants who have no prior exposure to a VR-based dementia education program. For this study, they will only receive the standard course material on dementia through the university's e-learning platform. They will not receive any ASA VR content.
  Purpose: This group acts as a true control, representing the outcomes of conventional dementia education through the university's regular e-learning, for students who have not had any previous VR exposure.
  Interventions: Other: VR-Unexposed + Standard Control Group

INTERVENTIONS:
Other: VR-Experienced + ASA VR Group — Participants will attend a single 60-minute session consisting of five components: a 5-minute introduction to welcome participants and outline objectives, followed by a 10-minute study briefing in which the PI explains the study aims, participant roles, and emphasizes voluntary participation, confidentiality, and informed consent. The core 30-minute intervention involves a scenario-driven Virtual Reality Dementia Game where participants role-play interactions with an AI avatar simulating a person living with dementia. The structured storyline is designed to immerse learners in realistic care situations, directly supporting the learning objectives while fostering empathy, understanding, and positive attitudes toward dementia care. Immediately after, students complete a 10-minute post-program questionnaire (T4) to assess attitudinal and knowledge changes. The session concludes with a 5-minute closing that summarizes the activities.
  Arms: VR-Experienced + ASA VR Group
Other: VR-Experienced + Standard Control Group — Participants in these arms will access dementia-related content through the university's existing e-learning platform as part of their regular curriculum. These groups will not receive a special intervention session from this study and will serve as control groups for the ASA VR program. All participant groups will complete the post-intervention (T4) questionnaires at designated times to measure the study's primary and secondary outcomes.
  Arms: VR-Experienced + Standard Control Group
Other: VR-Unexposed + ASA VR Group — Participants will attend a single 60-minute session consisting of five components: a 5-minute introduction to welcome participants and outline objectives, followed by a 10-minute study briefing in which the PI explains the study aims, participant roles, and emphasizes voluntary participation, confidentiality, and informed consent. The core 30-minute intervention involves a scenario-driven Virtual Reality Dementia Game where participants role-play interactions with an AI avatar simulating a person living with dementia. The structured storyline is designed to immerse learners in realistic care situations, directly supporting the learning objectives while fostering empathy, understanding, and positive attitudes toward dementia care. Immediately after, students complete a 10-minute post-program questionnaire (T4) to assess attitudinal and knowledge changes. The session concludes with a 5-minute closing that summarizes the activities.
  Arms: VR-Unexposed + ASA VR Group
Other: VR-Unexposed + Standard Control Group — Participants in these arms will access dementia-related content through the university's existing e-learning platform as part of their regular curriculum. These groups will not receive a special intervention session from this study and will serve as control groups for the ASA VR program. All participant groups will complete the post-intervention (T4) questionnaires at designated times to measure the study's primary and secondary outcomes.
  Arms: VR-Unexposed + Standard Control Group

SUMMARY:
•Terminology Clarification: In the previous study (NCT06629844), the term ' virtual reality (VR)' referred to a 360-degree video viewed through a VR headset. This format offered an immersive experience but was non-interactive. In contrast, the current study uses an 'ASA VR' intervention, which is a scenario-driven, interactive virtual reality simulation. Participants take part in role-playing with an artificial intelligence (AI) character representing a person living with dementia. This distinction is crucial for understanding the study design and results, as the cognitive and experiential demands of the two formats differ greatly.

•Brief Summary: This nested 2x2 factorial quasi-experimental design study focuses on Indonesian nursing students and aims to examine the effectiveness of scenario-driven virtual reality (VR) dementia educational programs. The study uses a four-arm design to evaluate different combinations of interventions.

The study addresses the following research questions:

What is the effect of a Scenario-Driven VR dementia education program on improving participants' attitude, knowledge, intention to help people living with dementia, ageist attitudes, and participant satisfaction with the Scenario-Driven VR dementia education program?

Participants will voluntarily join a 30-minute class education program, with each participant attending only once. The program, integrated into the faculty's dementia-related courses, will be structured around a series of components, including an introduction, Scenario-Driven VR, a post-program questionnaire, and a conclusion.

DETAILED DESCRIPTION:
•Detailed Description:

1. Research Implementation

   1. ASA Program Overview ASA VR is a scenario-driven, interactive virtual reality (VR) learning experience designed to cultivate dementia-competent attitudes and behaviors among healthcare students. Unlike the passive 360° video used in the prior study, ASA requires learners to make decisions, engage in role-play with an AI character portraying a person living with dementia (PLWD), and receive immediate, context-specific feedback.
   2. Educational Concept and Design Rationale ASA operationalizes evidence-informed instructional principles: (1) problem-centered, authentic tasks with demonstration and guided practice; (2) anchored, scenario-based learning to encourage transfer; and (3) first-person immersive perspective-taking shown to strengthen empathy in healthcare education using VR. Together, these elements aim to move learners beyond recognition-level knowledge to a situated judgment and prosocial intention.
2. Research Method This study is randomized with parallel assignment. study aims to evaluate scenario-driven VR dementia education programs among nursing students in Indonesia. The participants will be nursing students who are enrolled in specific semesters and courses designated for the implementation of this educational program. The study will be conducted with students in the sixth semester (third year). Participants in this study were drawn from the previous study (NCT06629844). The previous study was a quasi-experimental, two-arm design, consisting of an intervention group that received an education program using VR and a control group that attended conventional classes. In the previous study, we collected questionnaires at three time points: pre-questionnaire (T1), post-questionnaire (T2), and a follow-up questionnaire three months later (T3). In this study, we continue our research using the Scenario-Driven VR Dementia Education Program. We will conduct randomized with parallel assignment study with four arms. The intervention group from the previous study, who had prior VR experience, will be divided into two groups: one receiving the Scenario-Driven VR Dementia Education Program and one serving as a control group. Similarly, the control group from the previous study will also be divided into two groups: one receiving the Scenario-Driven VR Dementia Education Program and one serving as a control group. After finishing the Scenario-Driven VR Dementia Education Program, we will give a post-questionnaire (T4).

All prospective participants will be assigned new ID numbers to ensure the confidentiality of their student ID numbers. Each new ID will correspond to the participant's ID number from the previous study, with the addition of a code to classify them into four groups. This approach will allow us to link participant data in the current study with data from the previous study. The randomization will be perform using computer randomization. The protocol has been reviewed and approved by the Ethics Committee of the Faculty of Nursing, Universitas Airlangga. The Scenario-Driven VR dementia education program will not be integrated into a specific class, but will cover themes related to dementia care. Participants will be recruited through class announcements. An overview of the research process will be provided, and detailed instructions regarding the study will be given shortly before it begins. The research team will announce the study approximately one week in advance, and recruitment will be conducted via Google Forms. Students who register will be randomly assigned to four groups. Selected participants will receive their ID numbers along with details about the program's schedule and location through a class announcement three days prior to the intervention.

On the day of the intervention, participants will attend the designated location and sign an attendance sheet using their IDs. The Principal Investigator (PI) will explain the study's stages and emphasize that participants can withdraw at any time without any consequences. Participation in the study will be entirely voluntary, and there will be no coercion. Students who agree to participate in the study will provide informed consent. Those in the program will complete a questionnaire after the intervention. Regarding recruitment, eligible participants will be identified through the previous study's data. Students registered in the selected courses for the 2025/2026 academic year. All eligible students will receive comprehensive information about the study and an invitation to participate. Both the intervention and control groups will complete post-intervention questionnaires.

The intervention group will receive the Scenario-Driven VR Dementia Education Program, while the control group will attend an online class to receive information about the study, provide informed consent, and complete the post-test questionnaire. Both the intervention and control sessions will be conducted once. Students who provide informed consent in the intervention group will attend a classroom lecture to participate in the Scenario-Driven VR Dementia Education Program and then complete a post-lecture survey (T4). The control group will follow the same timeline for completing the survey (T4).

In the previous study, students experienced a non-interactive 360° video via a headset, which likely enhanced presence and baseline attitude but required no active problem-solving. In this follow-up study, we investigate whether ASA's interactivity provides incremental value (in the form of additive or synergistic effects) beyond prior passive immersion. This design allows us to disentangle (A) the main effect of ASA and (B) whether prior 360° exposure primes learners for greater gains when interactivity is introduced.

ELIGIBILITY:
Inclusion Criteria:

* Registered nursing students at Universitas Airlangga in the designated semester and courses (academic year 2025/2026).
* Provide informed consent.

Exclusion Criteria:

* Not enrolled in the specified semester/courses.
* Prior participation in a scenario-driven VR dementia education program similar to ASA VR that could influence outcomes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: Attitudes Toward People with Dementia Scale | Immediately post-intervention (T4), on the same day, within 0-60 minutes after session end.
  Participants' attitudes toward persons living with dementia (PLWD) will be assessed using the Attitudes Toward People with Dementia Scale, developed by Kim K and Kuroda K. (Kim K, Kuroda K. Factors related to attitudes toward people with dementia: Development of the Attitude Toward Dementia Scale and Dementia Knowledge Scale. Bulletin of Social Medicine. 2011; 28(1), 43-55). The original scale was published in Japanese, and a forward-backward translation process was conducted to produce the Indonesian version of the scale.
  The questionnaire consists of 14 items and is designed to evaluate participants' attitudes toward PLWD. The estimated time to complete the questionnaire is 3-5minutes.

SECONDARY OUTCOMES:
Knowledge of Dementia | Immediately post-intervention (T4), on the same day, within 0-60 minutes after session end.
  Participants' knowledge of dementia will be assessed using the Dementia Knowledge Scale, developed by Kim and Kuroda (2011). This scale was originally designed to measure various aspects of dementia knowledge, including symptoms, causes, progression, and caregiving strategies. The scale consists of 15 multiple-choice and true/false questions that cover a broad range of dementia-related topics. The Indonesian version of the scale was created through a forward-backward translation process to ensure cultural and linguistic accuracy. Higher scores on this scale indicate a better understanding of dementia
Intention to Help Persons Living with Dementia | Immediately post-intervention (T4), on the same day, within 0-60 minutes after session end.
  To assess participants' intention to help PLWD, we will use a set of four vignettes based on the study by Matsumoto et al. (2022). Each vignette presents a realistic scenario in which a person with dementia may need assistance, such as confusion in a public place, difficulty with daily tasks, or issues related to memory loss. Participants will read through each vignette and indicate their intended helping behavior on a 4-point Likert scale (ranging from "definitely would not help" to "definitely would help"). The vignettes are designed to assess the participants' willingness to offer practical, emotional, or social support to PLWD in everyday situations. The Indonesian version of the vignettes and Likert scale has also undergone a forward-backward translation to ensure that the language and context are appropriate for Indonesian nursing students.
Ageist Attitudes Towards Older Adults | Immediately post-intervention (T4), on the same day, within 0-60 minutes after session end.
  Participants' ageist attitudes will be assessed using selected items from the Fraboni Scale of Ageism (FSA). The FSA is a validated instrument developed by Fraboni et al. (1990) that measures stereotypes, prejudice, and discriminatory attitudes toward older adults. In this study, a subset of key items will be adapted and translated into Indonesian version using a forward-backward translation process to ensure cultural and linguistic appropriateness. The selected items cover three main domains: Stereotyping, Social distancing, Discriminatory attitudes. Each item will be rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), with higher scores indicating stronger ageist attitudes. This measure will allow researchers to explore how underlying biases may impact students' empathy, communication, and willingness to provide equitable dementia care to older adults.
User Experience Questionnaire | Immediately post-intervention (T4), on the same day, within 0-60 minutes after session end.
  To assess participants' perceptions of the VR dementia education program, we will use the User Experience Questionnaire (UEQ). This questionnaire evaluates users' experiences with the VR program across several dimensions, such as attractiveness, perspicuity, efficiency, dependability, stimulation, and novelty. The UEQ was used previously in similar studies and provides valuable feedback on the user experience. The Indonesian version of the UEQ, authored by Harry B. Santoso https://www.ueq-online.org/ , will be employed to ensure the questionnaire is culturally and linguistically appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Airlangga, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The IPD associated with participants' real IDs will be retained only by the PI of this study.
  New datasets will use new IDs so that only the PI can link the research data to participants' original IDs.
  Datasets that use the new IDs will be shared with the research team for data processing purposes (statistical analysis plan, SAP) and publication. All data will be stored for five years (September 2025- September 2030).
  Datasets will not be made public and will only be shared with the project's research team.

REFERENCES:
- [Background] Wu J, Igarashi A, Suzuki H, Matsumoto H, Kugai H, Takaoka M, Yamamoto-Mitani N. Effects of a dementia educational programme using virtual reality on nurses in an acute care hospital: A pre-post comparative study. Int J Older People Nurs. 2024 May;19(3):e12616. doi: 10.1111/opn.12616. PMID 38769648
- [Background] Suzuki H, Igarashi A, Matsumoto H, Kugai H, Takaoka M, Sakka M, Ito K, Hagiwara Y, Yamamoto-Mitani N. A Dementia-Friendly Educational Program Using Virtual Reality for the General Public in Japan: A Randomized Controlled Trial for DRIVE. Gerontologist. 2024 Nov 1;64(11):gnae113. doi: 10.1093/geront/gnae113. PMID 39140623
- [Background] Sari DW, Igarashi A, Takaoka M, Yamahana R, Noguchi-Watanabe M, Teramoto C, Yamamoto-Mitani N. Virtual reality program to develop dementia-friendly communities in Japan. Australas J Ageing. 2020 Sep;39(3):e352-e359. doi: 10.1111/ajag.12797. Epub 2020 Jun 2. PMID 32483931

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT07238439/Prot_SAP_ICF_000.pdf